CLINICAL TRIAL: NCT01126476
Title: Retreatment of Recurrent Tumors Using Proton Therapy
Brief Title: Proton Radiotherapy for Recurrent Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 23309
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Tumors
Keywords: Adults with non-CNS recurrent tumors who have been previously irradiated; and have a tumor recurrence in or near prior radiation fields
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- small volume strata (Active Comparator): 12 in small volume strata
  Interventions: Other: Proton Radiotherapy
- large volume strata (Active Comparator): 12 in large volume strata
  Interventions: Other: Proton Radiotherapy

INTERVENTIONS:
Other: Proton Radiotherapy

SUMMARY:
The purpose of this study is to determine the feasibility of using proton radiotherapy for reirradiation of recurrent malignancies.

DETAILED DESCRIPTION:
Patients will be stratified by treatment site (Head and Neck, Thorax, Abdomen, Pelvis, Extremities) and by treatment volume (low volume, high volume) for a total of 10 strata. This study will be done in two phases. In the first phase, feasibility will be established using the primary objectives set below. The second phase will begin no earlier than 90 days after the last patient in the initial phase has completed treatment in each strata and once feasibility has been verified. The secondary objectives will serve as the objectives for the second phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed, non-CNS solid malignancies who have been previously radiated and have a tumor recurrence in or near prior radiation fields. Re-biopsy of the recurrence is not required and left to the discretion of the treating physician, although every effort should be made to confirm recurrence.
* Patients must have a Karnofsky Performance Status of 60. Life expectancy of 3 months .
* Age greater or equal to 18.
* Patients must be able to provide informed consent.
* Women of child bearing potential as long as she agrees to use a recognized method of birth control (e.g. oral contraceptive, IUD, condoms or other barrier methods, etc.)
* Hysterectomy or menopause must be clinically documented.

Exclusion Criteria:

* Prior radiation treatment less than 3 months from planned start of re-irradiation of any part of the intended treatment volume.
* Pregnant women, women planning to become pregnant and women that are nursing.
* Actively being treated on any research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Feasibility of proton therapy | 90 days
  To determine if the study is infeasible, defined if greater than 10% of pts experience one of the following:
  1. Patient cannot be given treatment because anatomy is such that a dosimetrically satisfactory treatment plan cannot be devised.
  2. Patient who receives 15% or more of their treatments (for any reason, i.e. unable to set patient up within acceptable limits of tolerance, patient unable to tolerate treatment position or immobilization for duration of treatment) using photon radiotherapy (i.e. up to 15% of treatments could be delivered using photons).
  3. Patient is unable to complete all of his/her treatments within 10 days of estimated date of treatment completion or requires a treatment break greater than 5 days.
Acute Toxicity | within 90 days
  Acute Toxicity is defined as any grade 4 toxicity observed within 90 days from the initiation of radiotherapy that is felt to be directly related to their proton treatment. Toxicities will be graded by NCI CTC Version 4.0

SECONDARY OUTCOMES:
Late toxicity | open-ended
  Late toxicity is defined as any grade 3 or higher toxicity observed later than 90 days from start of therapy. Late toxicities will be graded according to the RTOG/EORTC late morbidity scoring system.

CONTACTS AND LOCATIONS:
Overall Officials: John Plastaras, MD, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine; Marcio Fagundes, MD, Principal Investigator — Procure, Oklahoma City, OK; William F. Hartsell, MD, Principal Investigator — ProCure Proton Therapy Center, Warrenville, IL
Locations (3):
- United States (3):
  - ProCure Proton Therapy Center, Warrenville, Illinois
  - Procure, Oklahoma City, Oklahoma
  - Abamson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania